CLINICAL TRIAL: NCT06587893
Title: Anatomical Observational Study of the Characteristics of the Suprascapular Notch Using Ultrasound.
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Pierre Goffin, Head of Acute Medicine department, University of Liege
Other Study IDs: Anatomie NSS
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Suprascapular Nerve Block
Keywords: anatomy; suprascapular notch; sono-anatomy; bones variations
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- healthy adult volunteer group: hospital workers recruited in intensive care and emergency departments.
  Interventions: Other: echography

INTERVENTIONS:
Other: echography — performance of ultrasound of the scapular regions to identify and measure the suprascapular notch in our group of healthy adult volunteers.

SUMMARY:
Carrying out an anatomical study to describe the suprascapular notch. The project is to determine the characteristics (measured dimensions and shapes) of the suprascapular notch by ultrasound measurements on a series of healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* all adult hospital workers from the two departments concerned

Exclusion Criteria:

* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
lenght | The ultrasound measurement will be carried out only once for each volunteer participant. The time spent participating in the study will be approximately 10 minutes per participant (time required for ultrasound measurements).
  Measuring the length and depth of the notch. Calculating the length/depth ratio. Measurements in millimeters.
  The measurement will be made on each side: left and right.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Goffin, MD MSc, Principal Investigator — Groupe Santé CHC - Liège - Belgium
Locations (1):
- MontLegia Hospital, Groupe Santé CHC, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided